CLINICAL TRIAL: NCT02701543
Title: Prospective, Randomized, Multi-Center Study for the Treatment of Subjects With Symptomatic Femoropopliteal Artery Disease With the Ranger Paclitaxel Coated PTA Balloon Catheter (Study Arm) Versus the IN.PACT Drug Eluting Balloon (Control Arm)
Brief Title: Compare I Pilot Study for the Treatment of Subjects With Symptomatic Femoropopliteal Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Dierk Scheinert, Prof. Dr., University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP_14/001
Record Dates: First submitted 2016-01-19; First posted 2016-03-08 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranger Drug Eluting Balloon (Active Comparator): Intervention with Over the Wire (OTW) Percutaneous transluminal angioplasty (PTA )balloon catheter with a semi-compliant balloon coated with a formulation of 2μg/mm2 paclitaxel and acetyl tri-n-butyl citrate (ATBC) as carrier substance
  Interventions: Device: Ranger Drug Eluting Balloon
- In Pact Drug Eluting Balloon (Active Comparator): Intervention with Over the Wire (OTW) peripheral balloon catheter. The balloon surface is coated with a formulation of 3μg/mm2 paclitaxel and urea as carrier substance.
  Interventions: Device: In Pact Drug Eluting Balloon

INTERVENTIONS:
Device: Ranger Drug Eluting Balloon — Percutaneous transluminal angioplasty (PTA), in which a balloon is advanced and inflated in the obstructed artery for several seconds to minutes, has become the standard endovascular treatment for peripheral arteries
  Arms: Ranger Drug Eluting Balloon
Device: In Pact Drug Eluting Balloon — Percutaneous transluminal angioplasty (PTA), in which a balloon is advanced and inflated in the obstructed artery for several seconds to minutes, has become the standard endovascular treatment for peripheral arteries
  Arms: In Pact Drug Eluting Balloon

SUMMARY:
To compare two different Paclitaxel coated balloons in the treatment of high grade stenotic or occluded lesions in Superficial femoropopliteal artery (SFA )and/or Proximal Popliteal Artery in Peripheral Artery Disease (PAD) patients with Rutherford class 2-4.

DETAILED DESCRIPTION:
This study is a prospective, multi-center 1:1 randomized trial. Patients will be stratified according to lesion length (≤ 10 cm/ > 10 cm and < 20 cm / > 20 cm and ≤ 30 cm). Each strata will include approximately 138 patients.

The trial is to investigate the safety and efficacy of the Ranger™ Drug Coated Balloon in comparison to the IN.PACT™ Drug Coated Balloon in patients with symptomatic femoropopliteal artery disease.

All enrolled subjects will be followed through to 24 months to assess the incidence of restenosis by ultrasound and major adverse events (MAE). Follow-up visits occur at 1, 6, 12 and 24-month intervals per local standard of care. Telephone follow-up visits will occur at 36, 48 and 60 month.

Up to 414 patients will be enrolled at approximately 10-18 sites in Germany for comparison between the following two groups:

Treatment with the Ranger™ Paclitaxel Coated Balloon Catheter (Boston Scientific Corporation, Natick, MA, USA) vs. the IN.PACT™ Drug Eluting Balloon (Medtronic Inc., Minneapolis, MI, USA).

ELIGIBILITY:
Inclusion Criteria:

1. Subject age ≥ 18
2. Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved consent form Subject understands the duration of the study, agrees to attend follow-up visits, and agrees to complete the required testing Rutherford category 2-4.
3. Subject has a de novo or restenotic lesion with ≥ 70% stenosis documented angiographically and no prior stent in the target lesion.
4. Target lesion length is ≤ 30cm
5. Target lesion is at least 1cm below the origin of the profunda femoris and does not exceed the medial femoral epicondyle.
6. Multiple lesions with max. 3cm healthy vessel segment in between lesions can be considered at the discretion of the operator as one lesion. Total lesion length should not exceed 30 cm.
7. Reference vessel diameter (RVD) ≥ 4 mm and ≤ 6.5 mm by visual estimation.
8. Patency of at least one (1) infrapopliteal artery to the ankle (< 50% diameter stenosis) in continuity with the native femoropopliteal artery.
9. A guidewire has successfully traversed the target treatment segment.

Exclusion Criteria:

1. Failure to successfully cross the target lesion
2. Angiographic evidence of severe calcification
3. Presence of fresh thrombus in the lesion.
4. Presence of aneurysm in the target vessel/s
5. Presence of a stent in the target lesion
6. Prior vascular surgery of the target lesion.
7. Stroke or heart attack within 3 months prior to enrollment
8. Any surgical procedure or intervention performed within 30 days prior to or post index procedure
9. Superficial femoropopliteal Artery or Proximal popliteal artery disease in the opposite leg that requires treatment at the index procedure
10. Target lesion requires treatment with alternative therapies such as stenting, laser, atherectomy, cryoplasty, brachytherapy, re-entry devices
11. Enrolled in another investigational drug, device or biologic study
12. Life expectancy of less than one year
13. Known allergies or sensitivity to heparin, aspirin, other anticoagulant/ antiplatelet therapies, paclitaxel or contrast media that cannot be adequately pre-treated prior to index procedure
14. Rutherford classification of 0, 1, 5 or 6.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Patency rate | 1 year
  Efficacy: patency rate after one year defined as absence of clinically driven Target Lesion Revascularization (due to symptoms and drop of ABI of ≥ 20% or > 0.15 when compared to post-procedure ) or restenosis with Peak Velocity Ratio > 2.4 evaluated by Duplex Ultrasound
Composite of freedom from device and procedure-related death through 12 months post procedure as well as freedom from both target limb major amputation and clinically-driven target vessel revascularization | 1 year
  Composite of freedom from device and procedure-related death through 12 months post procedure as well as freedom from both target limb major amputation and clinically-driven target vessel revascularization

SECONDARY OUTCOMES:
Target Lesion Revascularization (TLR) rate | 6,12,24 months
  Target Lesion Revascularization rate at 6, 12, 24, 36, 48 and 60 months
Walking capacity | 6,12,24 months
  Walking capacity assessment by Walking Impairment Questionnaire (WIQ) at 6, 12 and 24 months versus baseline.
binary restenosis | 6,12,24 months
  Duplex-defined binary restenosis (Peak systolic velocity ratio >2.4) of the target lesion post-procedure and at 6, 12 and 24 months or at any time of re-intervention
improvement shift in Rutherford classification | 6,12,24 months
  Sustained clinical improvement: an improvement shift in the Rutherford classification of one class in amputation and Target Vessel Revascularization free surviving patients at 12 months
secondary Safety | 60 months
  Composite of freedom from device and procedure-related death through 60 months post procedure as well as freedom from both target limb major amputation and clinically-driven target vessel revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Dierk Scheinert, Prof.Dr., Principal Investigator — University Leipzig
Locations (1):
- University Clinic Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Steiner S, Schmidt A, Zeller T, Tepe G, Thieme M, Maiwald L, Schroder H, Euringer W, Popescu C, Brechtel K, Brucks S, Blessing E, Schuster J, Langhoff R, Schellong S, Weiss N, Beschorner U, Wittig T, Scheinert D. Low-Dose vs High-Dose Paclitaxel-Coated Balloons for Femoropopliteal Lesions: 2-Year Results From the COMPARE Trial. JACC Cardiovasc Interv. 2022 Oct 24;15(20):2093-2102. doi: 10.1016/j.jcin.2022.08.004. Epub 2022 Sep 28. PMID 36265942
- [Derived] Steiner S, Schmidt A, Zeller T, Tepe G, Thieme M, Maiwald L, Schroder H, Euringer W, Ulrich M, Brechtel K, Brucks S, Blessing E, Schuster J, Langhoff R, Schellong S, Weiss N, Scheinert D. COMPARE: prospective, randomized, non-inferiority trial of high- vs. low-dose paclitaxel drug-coated balloons for femoropopliteal interventions. Eur Heart J. 2020 Jul 14;41(27):2541-2552. doi: 10.1093/eurheartj/ehaa049. PMID 31989155